CLINICAL TRIAL: NCT05366504
Title: Is Combined Low Intensity Shockwave Therapy (LiST) Plus Platelet-rich Plasma (PRP) Injection Therapy Better Than LiST Monotherapy for the Improvement of Erectile Function? a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: LiST Plus PRP Injection Therapy vs LiST Monotherapy for ED Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases Theesaloniki, Greece, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMOP
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Combination Product: LiST + PRP intracorporeal injection
- Group B (Placebo Comparator)
  Interventions: Combination Product: LiST + Placebo(normal saline intracorporeal injection)

INTERVENTIONS:
Combination Product: LiST + PRP intracorporeal injection — 12 LiST sessions (2 sessions per week) plus PRP (2 intracorporeal injections 3 weeks apart, after the 1st and the 7th LiST sessions) ( 30 patients).
  Arms: Group A
Combination Product: LiST + Placebo(normal saline intracorporeal injection) — All subjects of this group will receive 12 sessions (V3-V14) of LiST with session frequency 2/week and 2 normal saline injections with 3 weeks treatment interval (V3 and V9), 10 ml of normal saline will be injected at each session.
  Arms: Group B

SUMMARY:
We designed a double blind randomized sham-controlled trial in order to investigate and compare the treatment efficacy of LiST plus PRP intracorporeal injection vs LiST plus placebo (normal saline intracorporeal injection) in men with moderate and mild to moderate vasculogenic ED, as measured by IIEF-EF.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 40-70 years.
3. Sexually active in a stable, heterosexual relationship of more than three months duration.
4. Presence of vasculogenic ED for at least 6 months.
5. IIEF-ED: 11-21 at visit 2
6. PDE5i users and report some/good response to PDE5i ( 5 points drop in the IIEF-ED after PDE5i wash-out) at the last month before screening.
7. Agree to suspend all ED therapy for the duration of the study.
8. Agree to attempt sexual intercourse at least 4 times every 4 weeks, for the duration of the study without being under the influence of alcohol or recreational drugs. Agree to document the outcome using the Sexual Encounter Profile (SEP) diary, as needed.

Exclusion Criteria:.

1. Previous major pelvic surgery or pelvic trauma that could impact erectile function, such as radical prostatectomy, radical cystectomy, rectal surgery. Patients with previous TURP surgery without sequelae of iatrogenic ED, may be included.
2. Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, grafting.
3. Previous history of priapism or penile fracture
4. Previous radiation therapy to pelvis.
5. Abnormal morning serum testosterone level defined as a value lower than 300 ng/dL (indicative of untreated hypogonadism), or greater than 1197 ng/dL.
6. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
7. Psychogenic ED.
8. Peyronie's Disease or penile curvature that negatively influences sexual activity.
9. Anatomical or neurological abnormalities in the treatment area.
10. Any untreated medical condition (medical history)
11. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's Disease.
12. Refusal to suspend ED therapy for duration of study. Subjects who are using Tadalafil as a treatment for BPH (Benign Prostatic Hyperplasia) will also be excluded.
13. Men deemed not healthy enough to participate in sexual activity.
14. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
15. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
16. History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
17. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using SSRI or psychotropic medications.
18. Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.
19. Patients with any hematological disorder.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the change of the IIEF-ED score from baseline to 4 weeks after final treatment | baseline and 4 weeks follow up visit
  EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction).

SECONDARY OUTCOMES:
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the change of the IIEF-ED score from baseline to 12 weeks after final treatment | baseline and 12 weeks follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the % of patients who attain MCID in IIEF-EF domain from baseline to 4 weeks after final treatment. | at 4 weeks follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED at baseline and by 2 or more in the EF domain score of the IIEF for patients with moderate ED at baseline
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the % of patients who attain MCID in IIEF-EF domain from baseline to 12 weeks after final treatment. | at 12 weeks follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED at baseline and by 2 or more in the EF domain score of the IIEF for patients with moderate ED at baseline
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the change of Sexual Encounter Profile Question 3 (SEP3) %Yes score from baseline to 4 weeks after final treatment. | baseline and 4 weeks follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
The difference between the LiST plus PRP injection group and the LiST plus normal saline injection group in the change of Sexual Encounter Profile Question 3 (SEP3) %Yes score from baseline to 12 weeks after final treatment. | baseline and 12 weeks follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
Number of patients with treatment related adverse events | 28 weeks
  Potential treatment related adverse events after the first treatment session and during the 3 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Professor, Principal Investigator — G.Gennimatas General Hospital, Thessaloniki,Greece

IPD SHARING:
Plan to Share IPD: No